CLINICAL TRIAL: NCT03544931
Title: The Impact of Enamel Matrix Derivatives on Markers of Systemic Inflammation After Flapless Periodontal Therapy
Brief Title: Enamel Matrix Derivatives on Systemic Inflammation After Periodontal Therapy
Acronym: PERIOEMD-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3649/15B
Record Dates: First submitted 2018-04-30; First posted 2018-06-04 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root Instrumentation + EMD Application (Experimental): Periodontal treatment is delivered with ultrasonic instrumentation performed with fine tips. The approach chosen is the one-stage full-mouth ultrasonic debridement in which all the treatment of diseased sites is performed within one hour.
  In this group, at the end of the instrumentation enamel matrix derivatives is placed in all sites with a periodontal pocket depth deeper than 5mm.
  Interventions: Procedure: Root Instrumentation; Device: EMD Application
- Root Instrumentation (Active Comparator): Periodontal treatment is delivered with ultrasonic instrumentation performed with fine tips. The approach chosen is the one-stage full-mouth ultrasonic debridement in which all the treatment of diseased sites is performed within one hour.
  Interventions: Procedure: Root Instrumentation

INTERVENTIONS:
Procedure: Root Instrumentation — Instrumentation of the root surface in order to achieve debridement
Device: EMD Application — Application of Enamel Matrix Derivatives on the root surface after debridement in sites with probing depth deeper than 5 mm
  Arms: Root Instrumentation + EMD Application

SUMMARY:
The aim of this study is to compare periodontal treatment with or without the adjunct of an enamel matrix derivative in terms of acute-phase responses in healthy patients.

DETAILED DESCRIPTION:
Patients with periodontitis will be randomly allocated to two groups. In both groups, periodontal root instrumentation will be performed. In the test group, an additional flapless application of enamel matrix derivatives will be granted for sites with pockets deeper than 5 mm.

Systemic inflammation as measured through blood testing and local parameters of periodontal health will be measured at baseline and three months after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* No previous periodontal treatment
* Presence of Periodontitis (Clinical attachment loss of at least 3 mm in 2 or more non-adjacent teeth)
* Ability to understand the study procedures and comply with them through the length of the study

Exclusion Criteria:

* Pregnancy and breast feeding
* Need for antibiotic treatment during periodontal therapy
* Chronic infections
* Systemic diseases
* Patients who report current smoking over 20 cigarettes per day

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change of C Reactive Protein (CRP) at 24 hour | Collected at Baseline and 24 hours in order to calculate the changes
  CRP analyzed though blood sampling. Unit of measure: mg/L

SECONDARY OUTCOMES:
Glucose | Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
Cholesterol | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
LDL Cholesterol | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
HDL Cholesterol | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
Triglyceride | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
Fibrinogen | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
D-Dimer | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/L
Cystatin C | Collected at Baseline, 24 hours and 3 months after treatment
  analyzed though blood sampling. Unit of measure: mg/L
Full-mouth plaque score (FMPS) | Measured at Baseline and 3 months after treatment
  Changes in Full-mouth plaque score, measuring the amount of dental plaque on the teeth orally through clinical examination. Unit of measure %. The scale ranges from 0% ( minimum value, i.e. plaque absent) to 100% ( maximum value: all areas are occupied by plaque). 0% would the ideal value. No sub-scales are included.
Full-mouth bleeding score (FMBS) | Measured at Baseline and 3 months after treatment
  Changes of Full-mouth bleeding score, measuring the number of gingival areas that bleed after gingival probe passage. It is measured orally through clinical examination. Unit of measure %. The scale ranges from 0% ( minimum value, i.e. gingival inflammation is absent) to 100% ( maximum value: all gingival areas are inflamed). 0% would the ideal value. No sub-scales are included.
Pocket probing depth (PPD) | Measured at Baseline and 3 months after treatment
  Changes in PPD , measured orally through clinical examination. Unit of measure: mm
Clinical attachment level (CAL) | Measured at Baseline and 3 months after treatment
  Changes in CAL , measured orally through clinical examination. Unit of measure: mm
Recession of the gingival margin (REC) | Measured at Baseline and 3 months after treatment
  Changes in REC, measured orally through clinical examination. Unit of measure: mm
Number of sites with Pocket probing depth deeper than 3mm | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: N
Number of sites with Pocket probing depth deeper than 5mm | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: N
Percentage of sites with Pocket probing depth deeper than 3mm | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: %
Percentage of sites with Pocket probing depth deeper than 5mm | Measured at Baseline and 3 months after treatment
  Changes, measured orally through clinical examination. Unit of measure: %
Percentage of bleeding sites which measured Pocket probing depth deeper than 5mm at baseline | Measured at Baseline and 3 months after treatment
  Changes , measured orally through clinical examination. Unit of measure: %
Number of bleeding sites which measured Pocket probing depth deeper than 5mm at baseline | Measured at Baseline and 3 months after treatment
  Changes , measured orally through clinical examination. Unit of measure: N
C Reactive Protein (CRP) at 3 months | Collected 3 months after treatment
  CRP analyzed though blood sampling. Unit of measure: mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Graziani F, Gennai S, Petrini M, Bettini L, Tonetti M. Enamel matrix derivative stabilizes blood clot and improves clinical healing in deep pockets after flapless periodontal therapy: A Randomized Clinical Trial. J Clin Periodontol. 2019 Feb;46(2):231-240. doi: 10.1111/jcpe.13074. PMID 30663788